CLINICAL TRIAL: NCT06062940
Title: SHARE Approach Evaluation
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 19-3053
Record Dates: First submitted 2023-09-07; First posted 2023-10-02 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Shared Decision Making

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Care Practice: We recruited 10 primary care practices from across Colorado, from all regions of the state (e.g., Eastern Plains, Mountain West, Front Range), and a mix of rural and urban practices of varying sizes. We recruited both practice staff and patients for this cohort.
  Interventions: Behavioral: SHARE Approach
- Cardiology Practice: We recruited 2 cardiology practices from across Colorado, from all regions of the state (e.g., Eastern Plains, Mountain West, Front Range), and a mix of rural and urban practices of varying sizes. We recruited both practice staff and patients for this cohort.
  Interventions: Behavioral: SHARE Approach

INTERVENTIONS:
Behavioral: SHARE Approach — The SHARE Approach training was given at each of these centers, teaching skills to clinicians about shared decision making.

SUMMARY:
The SHARE Approach Evaluation study was meant to evaluate the SHARE Approach, designed by AHRQ and updated by UCD. The SHARE Approach is a training program for clinicians on shared decision making.

DETAILED DESCRIPTION:
This research group has been selected by the Agency for Healthcare Research and Quality (AHRQ) to evaluate its SHARE Approach Model. This model is designed to improve shared-decision making (SDM) between providers and patients, and teaches clinicians skills that are applicable to SDM in the context of preference-sensitive treatment choice and problem-solving. It remains one of the only freely available SDM toolkits that provides clinician-facing resources for comprehensive SDM training. This study will assess the effectiveness of the SHARE model training using training evaluation surveys, card survey data with providers who have received the SHARE training, and their patients, and audio recordings of clinician/patient encounters. The training and evaluations will be done at a total of 12 health care practices (10 primary care practices and 2 cardiology practices). All research data will be de-identified and kept confidential.

ELIGIBILITY:
Inclusion Criteria:

* Population to be enrolled include clinicians and any practice staff who participate in the SHARE Approach training in 12 practices to be recruited across Colorado.
* Patients will also be enrolled for the card surveys and audio recordings if they are meeting with a clinician who has taken the SHARE Approach training.
* 18 to 89 years old

Exclusion Criteria:

* Children
* Decisionally challenged
* Prisoners

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Population to be enrolled include clinicians and any practice staff who participate in the SHARE Approach training in 12 practices to be recruited across Colorado.
  Patients will also be enrolled for the card surveys and audio recordings if they are meeting with a clinician who has taken the SHARE Approach training.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Clinician training evaluation: Confidence in ability to do shared decision making | pre-training, post-training, 2-month follow-up
  Clinician confidence in doing shared decision making was measured by a brief card survey question with a 5 point Likert scale. Possible scores range from 1 to 5, with lower scores indicating less usefulness and higher scores indicating more usefulness.
Clinician training evaluation: Confidence in understanding what shared decision making is | pre-training, post-training
  Clinician confidence in understanding shared decision making was measured by a brief card survey question with a 5 point Likert scale. Possible scores range from 1 to 5, with lower scores indicating less usefulness and higher scores indicating more usefulness.
Card survey: Clinician satisfaction with encounter | pre-training, 1 month post-training, 6 month follow-up
  Clinician satisfaction with encounter was measured by a brief card survey question with a 5 point Likert scale. Possible scores range from 1 to 5, with lower scores indicating less usefulness and higher scores indicating more usefulness.
Card survey: Patient satisfaction with encounter | pre-training, 1 month post-training, 6 month follow-up
  Patient satisfaction with encounter was measured by a brief card survey question with a 5 point Likert scale. Possible scores range from 1 to 5, with lower scores indicating less usefulness and higher scores indicating more usefulness.
Card survey: Clinician shared decision making (self-reported) | pre-training, 1 month post-training, 6 month follow-up
  After clinician/patient encounters, clinicians were asked to fill out a brief card survey rating shared decision making that occurred during the encounter. These include questions from the Dyadic OPTION (observing patient involvement in decision making) scale. Higher scores reflected better experiences of shared decision making, whereas lower scores reflected poorer experiences of shared decision making.
Card survey: Patient shared decision making (self-reported) | pre-training, 1 month post-training, 6 month follow-up
  After clinician/patient encounters, patients were asked to fill out a brief card survey rating their experiences with shared decision making during the encounter. These included questions modified from the Dyadic OPTION (observing patient involvement in decision making) scale. Higher scores reflected better experiences of shared decision making, whereas lower scores reflected poorer experiences of shared decision making.
Audio recordings: Shared Decision Making (highest score of topics discussed) | pre-training, 1 month post-training, 6 month follow-up
  A subset of clinician/patient encounters were audio recorded, and then coded using a modified OPTION (observing patient involvement in decision making) 12 coding schema for elements of shared decision making occurring within the encounter. As a primary outcome, we selected the highest-scored topic discussed in each encounter. Higher scores reflected better experiences of shared decision making, whereas lower scores reflected poorer experiences of shared decision making.
Clinician training evaluation: Overall evaluation of the SHARE training | post-training
  clinicians answered the question: Overall, what was your experience of the training you received today. Likert rating scale was "Very positive" to "Very negative"

SECONDARY OUTCOMES:
Shared Decision Making (total score) | pre-training, 1 month post-training, 6 month follow-up
  Clinician/patient encounters were audio recorded, and then coded using a modified OPTION (observing patient involvement in decision making) 12 coding schema for different elements of shared decision making within the encounter.
  The secondary outcome was the total score for each encounter, which averaged across scores for all topics discussed. Higher scores reflected better experiences of shared decision making, whereas lower scores reflected poorer experiences of shared decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Scherer, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No